CLINICAL TRIAL: NCT02076438
Title: Probiotics for Prevention of Antibiotic Associated Diarrhea and Clostridium Difficile Associated Disease in Hospitalized Adults-A Double Blind Placebo Controlled Trial
Brief Title: Probiotics for Prevention of Antibiotic Associated Diarrhea and Clostridium Difficile Associated Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Saint Peters University Hospital (Other)
Responsible Party: Principal Investigator, Amita Avadhani, DNP, DCC, ACNP, ANP, CCRN, Assistant Professor/Director Post MSN-DNP program, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro2012002450; Grant# PC 14-13 (Other: New Jersey Health Foundation)
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diarrhea
Keywords: antibiotics; diarrhea; c diff; Hospitalized patients
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: Probiotics
- Probiotics (Experimental): Lactobacillus Rhamnosus GG 10 billion cfu BID
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Randomized to receive probiotics or placebo
  Other Names: Lactobacillus Rhamnosus GG 10 billion cfu bid

SUMMARY:
The study will evaluate if administration of probiotic Culturelle (Lactobacillus Rhamnosus GG) along with antibiotics can help decrease the occurrence of diarrhea caused by antibiotics as well as Clostridium difficile Diarrhea.

DETAILED DESCRIPTION:
Inpatient adult males and females who are at least 18 years of age or older, undergoing treatment with antibiotics irrespective of indication and the type of antibiotics. The setting is an academic hospital.The patients are screened and potentially recruited upon initiation of antibiotic treatment regardless of indication for antibiotic prescription. The participants are patients being admitted to any inpatient units of the hospital for treatment with antibiotics. Exclusion criteria is:

* Diarrhea on admission or within the preceding week
* Reported recurrent diarrhea
* Bowel pathology that could result in diarrhea (including preexisting Inflammatory Bowel disease{IBD}, all forms for colitis or any other condition resulting in preexisting diarrhea)
* Intake of high risk antibiotics (clindamycin, cephalosporins, aminopenicillins→ well known to cause CDAD) and or more than two courses of other antibiotics in the past four weeks to exclude pre-existing diarrhea associated with antibiotic use
* Immunosuppression (Chronic steroid use, Active chemotherapy, Active radiotherapy, HIV or any other disorder resulting in a compromise in participants immune status)
* Bowel surgery causing liquid stools
* Regular probiotic intake before admission
* Lactose intolerance or intolerance to dairy products.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient adult males and females who are at least 18-89 years of age, undergoing treatment with antibiotics irrespective of indication and the type of antibiotics.

Exclusion Criteria:

* Diarrhea on admission or within the preceding week
* Reported recurrent diarrhea
* Bowel pathology that could result in diarrhea (including preexisting Inflammatory Bowel disease{IBD}, all forms for colitis or any other condition resulting in preexisting diarrhea)
* Intake of high risk antibiotics (clindamycin, cephalosporins, aminopenicillins→ well known to cause CDAD) and or more than two courses of other antibiotics in the past four weeks to exclude pre-existing diarrhea associated with antibiotic use
* Immunosuppression (Chronic steroid use, Active chemotherapy, Active radiotherapy, HIV or any other disorder resulting in a compromise in participants immune status)
* Bowel surgery causing liquid stools
* Regular probiotic intake before admission
* Lactose intolerance or intolerance to dairy products

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diarrhea | 4 weeks
  Diarrhea associated with antibiotics

SECONDARY OUTCOMES:
Tolerability of probiotics | 4 weeks
  Patient experience with use of probiotics

CONTACTS AND LOCATIONS:
Overall Officials: Amita Avadhani, DNP, Principal Investigator — Rutgers University and Saint Peters University Hospital
Locations (1):
- Saint Peters University Hospital, New Brunswick, New Jersey, United States